CLINICAL TRIAL: NCT05206097
Title: Determinants of Daily Physical Activity Level in Patients With Cystic Fibrosis - Pilot Study. Protocol
Brief Title: Determinants of Daily Physical Activity Level in Patients With Cystic Fibrosis - Pilot Study Protocol
Acronym: APM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 87RI20_0010 (APM)
Record Dates: First submitted 2022-01-10; First posted 2022-01-25 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; barriers and facilitators; daily physical activity; accelerometry
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity Program (Experimental)
  Interventions: Device: Accelerometer

INTERVENTIONS:
Device: Accelerometer — For the following study, each patient will be asked to wear a portable device over a 7-day period. The accelerometer will be previously set up according to anthropometric data of the patient and scheduled to automatically start and stop accelerations registration. The patient will be asked to wear the sensor as frequently as possible, with the exception of sleep period and during aquatic activities. A diary will be delivered to the patient in order to notify any problem/issue observed during the evaluation week (for example forgetting to wear the sensor). The accelerometry assessment will be associated to a questionnaire. Each patient will have to fill in it during the evaluation week. The questionnaire is composed of various questions from three different questionnaires: Ricci & Gagnon for subjective evaluation of PA level, CFQ-14+ for the evaluation of quality of life specifically in CF and EQ-5D for a more generic evaluation of quality of life.

SUMMARY:
The aim of the study is to analyze the determinants (barriers and facilitators) of the daily physical activity level in a population of patients with cystic fibrosis. A population of patients will be included in order to realize an assessment of their daily physical activity level over an entire week. A specific questionnaire, designed from 3 different questionnaires, will be associated to the physical activity evaluation and will allow to asses psycho-social and environmental factors.

DETAILED DESCRIPTION:
Physical activity (PA) is a major component of the management of patients with cystic fibrosis (CF). Regular PA is associated, in cystic fibrosis as in other pathologies, with health benefits and a greater life expectancy. However, the literature shows an absence of consensus for the daily PA level reached by CF patients, and also for the determinants of this PA level. It appears that CF patients tend to have a reduced PA level, compared to international guidelines. Some determinants have already been mentioned, like physical, psychological or organizational factors. But these factors have not been considered in a multifactorial way, by also considering social and environmental factors, and are rarely associated with objective PA level measurement or only reported in paediatric population. A better comprehension of these determinants of daily PA level represents an important issue for the optimization of interventions designed for the promotion of PA in cystic fibrosis.

For this study, a population of CF patients will realize an evaluation of their daily PA level based on accelerometry (by wearing a portable device over 7 days). During the PA assessment, patients will have a questionnaire to fill in, delivered with the sensor. The objective assessment of PA level will be analyzed with regard to various parameters from different dimensions: individual, clinical, psycho-social and environmental. Individual and clinical parameters will be collected from patients' data routinely assessed for the management of patients. Psycho-social and environmental parameters will be assessed with a specific questionnaire, specifically designed from 3 different questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis confirmed by the identification of genetic mutation and/or positive sweat test
* regular follow-up in CF centers ;
* age higher than 6 years old
* stable clinical status, away from exacerbation period or antibiotic treatment.

Exclusion Criteria:

* transplant patient or patient waiting for a transplant
* inability to fill in the questionnaire or to complete the planned evaluations
* ongoing participation in another research protocol (interventional study)
* refusal to participate in the study
* patient under legal protection.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Physical Activity Time | Week 1
  mean value of moderate to vigorous Physical Activity (MVPA) time (min/day), from an accelerometry evaluation over an entire week

SECONDARY OUTCOMES:
Daily Physical Activity level | Week 1
  Daily Physical Activity level, from the accelerometry evaluation compared to international PA guidelines
Duration of Physical Activity | Week 1
  Duration of Physical Activity performed by patients
Frequency of Physical Activity | Week 1
  Frequency of Physical Activity performed by patients
Type of Physical Activity | Week 1
  Type of Physical Activity performed by patients
Sedentarity time | Week 1
  Sedentarity time, from the accelerometry evaluation.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU DE BORDEAUX Hôpital des Enfants-Pellegrin - CRCM Pédiatrique, Bordeaux
  - CHU DE BORDEAUX Hôpital Haut-Lévêque - CRCM Adulte, Bordeaux
  - CHU DE LIMOGES Hôpital Dupuytren 2 - CRCM Adulte, Limoges
  - CHU DE LIMOGES Hôpital Mère Enfant - CRCM Pédiatrique, Limoges
  - CHU DE TOULOUSE Hôpital des Enfants - CRCM Pédiatrique, Toulouse
  - CHU DE TOULOUSE Hôpital Larrey - CRCM Adulte, Toulouse